CLINICAL TRIAL: NCT03096236
Title: Endoscopic Full-thickness Resection of Gastric Subepithelial Tumors With the gFTRD
Acronym: RESET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kliniken Ludwigsburg-Bietigheim gGmbH (Other)
Responsible Party: Sponsor
Other Study IDs: RESET
Record Dates: First submitted 2017-03-23; First posted 2017-03-30 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Feasibility, Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: EFTR — EFTR with the FTRD developed for gastric resection (gFTRD).

SUMMARY:
Subepithelial gastric tumors are rare and usually detected incidentally. Most subepithelial tumors (SET) are benign but up to 13% of all lesions can be malignant. Histology after needle biopsy often brings no clear diagnosis in SET, so further strategy often remains unclear. Surveillance endoscopy can be associated with the risk of progression. Endoscopic resection usually is difficult, associated with high risk of complications and sometimes is not feasible. Surgical resection is also associated with a risk of complications and often refused by the patients. With the developement of the gFTRD-System gastric SET can now be resected endoscopically. The advantage of this technique is the complete resection and a full-thickness resections specimen for are definite histology.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Gastric SET up to 15 mm (measurement: endoscopic ultrasound)

Exclusion Criteria:

* Age < 18 years
* Gastric SET > 15 mm and/or large extramural part
* Criteria of Lipoma (endoscopic ultrasound)
* Positive lymph nodes (endoscopic ultrasound)
* Stenosis (Esophagus)
* Diverticulum (Esophagus)
* Pregnancy or Nursing period

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastric SET
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Technical success | 1 minute (immediate)
  Successful enbloc- and macroscopically complete resection

SECONDARY OUTCOMES:
R0-Resection | three days
  Histologically confirmed complete resection
Histologically confirmed full thickness resection | three days
  Histologically confirmed full thickness resection
Procedure-associated complications | three months
  Procedure-associated complications such as bleeding or perforation
Necessity of surgical treatment | three months
  Necessity of surgical treatment
Residual or recurrent adenoma/carcinoma at endoscopic follow up | three months
  Residual or recurrent adenoma/carcinoma at endoscopic follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Ludwigsburg, Ludwigsburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meier B, Schmidt A, Glaser N, Meining A, Walter B, Wannhoff A, Riecken B, Caca K. Endoscopic full-thickness resection of gastric subepithelial tumors with the gFTRD-system: a prospective pilot study (RESET trial). Surg Endosc. 2020 Feb;34(2):853-860. doi: 10.1007/s00464-019-06839-2. Epub 2019 Jun 11. PMID 31187233